CLINICAL TRIAL: NCT01373385
Title: Prospective Pediatric Vesicoureteral Reflux Surgery Database
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Christina Kim, MD, Attending physician, Connecticut Children's Medical Center
Other Study IDs: 10-049
Record Dates: First submitted 2010-07-14; First posted 2011-06-15 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Vesicoureteral Reflux
Keywords: pediatric urology; vesicoureteral reflux; ureteral reimplant; Deflux
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical: Patients receiving a surgical procedure for vesicoureteral reflux at Connecticut Children's Medical Center.

SUMMARY:
The purpose of this research is to provide a clearer understanding of quality and outcomes for three types of surgical procedures performed at Connecticut Children's for treatment of vesicoureteral reflux. In order to consistently gather data over time, the investigators propose to establish database for surgical intervention for vesicoureteral reflux.

Specific Aim 1: To consistently collect performance and outcomes data for the surgical treatment of vesicoureteral reflux in order to increase internal understanding of these procedures.

Specific Aim2: To consistently collect performance and outcomes data for the surgical treatment of vesicoureteral reflux in order to perform more valuable clinical analysis for publication.

ELIGIBILITY:
Inclusion Criteria:

* Subject scheduled to receive surgical intervention for the treatment of vesicoureteral reflux at Connecticut Children's.

Exclusion Criteria:

* Subject not scheduled to receive surgical intervention for the treatment of vesicoureteral reflux at Connecticut Children's.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients receiving a surgical procedure for viesicoureteral reflux at Connecticut Children's Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2010-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Resolution of vesicoureteral reflux | Date of surgical intervention (day 1) to resolution of vesicoureteral reflux or additional surgical interventions for correction of vesicoureteral reflux, whichever comes first, or until enrollee's 18th birthday.
  Resolution of vesicoureteral reflux

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kim, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No